CLINICAL TRIAL: NCT05221684
Title: Lymph Node Ratio as a Predictor for Outcome in Rectal Cancer: a Retrospective Cohort
Brief Title: Lymph Node Ratio as a Predictor for Outcome in Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mostafa shalaby, MD, MSc, PhD, Lecturer of Colorectal Surgery, Mansoura University
Other Study IDs: LN ratio in rectal cancer
Record Dates: First submitted 2022-01-23; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Recurrence
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Lymph node harvesting — Lymph node harvesting after radical resection for rectal cancer with curative intent

SUMMARY:
This study aims to evaluate the value of the LNR as a prognostic indicator in patients with rectal cancer who offered total mesorectal excision.

DETAILED DESCRIPTION:
Patients and methods Study design and setting This is a retrospective review of prospectively collected and maintained database of patients with CRC admitted in the Oncology Center of Mansoura University (OCMU), the Colorectal Surgery Unit of Mansoura University Hospitals, and the Department of General Surgery of Alexandria University.

Selection criteria Patients of either gender aged 18 years or above who presented with rectal cancer of any stage will be included in the study. We will exclude patients with patients younger than 18 years; patients with synchronous colon cancer; synchronous liver, pulmonary or bones metastasis; or synchronous gastrointestinal cancer; or patients who were lost to follow-up.

Study endpoints The primary endpoint of the study is to assess the value of lymph node ratio (LNR) on the oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* rectal cancer of TNM stage I-III
* underwent radical resection with curative intent

Exclusion Criteria:

* synchronous colon cancer
* synchronous gastrointestinal cancer
* underwent palliative resection
* presented with intestinal obstruction
* those lost to follow-up.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with rectal cancer TNM stage I-III Who underwent surgery with curative intent
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-09 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Lymph node value | one year
  Value in prediction of oncological outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Shalaby, Principal Investigator — Mansoura Faculty of Medicine
Locations (1):
- Mansoura Faculty of Medicine, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided